CLINICAL TRIAL: NCT03768037
Title: A Study to Evaluate the Efficacy and Safety of Anlotinib Plus Pemetrexed as the 1-line Treatment of Patients With Platinum Intolerant Advanced Non-squamous NSCLC, With Pemetrexed Control.
Brief Title: Anlotinib Plus Pemetrexed or Pemetrexed for Previously Untreated Elderly (>=70) or PS=2 Non-squamous NSCLC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG1801
Record Dates: First submitted 2018-11-30; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-11

CONDITIONS: Advanced Non-squamous NSCLC
MeSH Terms: interventions — anlotinib; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib plus Pemetrexed (Experimental): Anlotinib plus Pemetrexed
  Interventions: Drug: Anlotinib plus Pemetrexed
- Pemetrexed (Other): Pemetrexed
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Anlotinib plus Pemetrexed — Anlotinib p.o, qd and it should be continued until disease progress or unacceptable toxic effects.
  Pemetrexed 500 mg/m2 every 21 days for 4-6 cycles or unacceptable toxic effects
  Arms: Anlotinib plus Pemetrexed
Drug: Pemetrexed — Pemetrexed 500 mg/m2 every 21 days for 4-6 cycles or unacceptable toxic effects
  Arms: Pemetrexed

SUMMARY:
Evaluate the efficacy and safety of Anlotinib plus Pemetrexed as the 1-line treatment of patients with Platinum intolerant advanced non-squamous NSCLC, with Pemetrexed control.

DETAILED DESCRIPTION:
Anlotinib (AL3818) is a kind of innovative medicines approved by State Food and Drug Administration（SFDA:2011L00661） which was researched by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd. Anlotinib is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR1、VEGFR2、VEGFR3、FGFR1/2/3、PDGFRa/β c-Kit and MET.

ELIGIBILITY:
Inclusion Criteria:

* ≥70 years old and ECOG PS=0-2 or ≥18 years old and ECOG PS=2
* Diagnosed with advanced or recurrent non-squamous NSCLC (phase IIIB/IV) through pathology, with measurable nidus(using RECIST 1.1)
* No prior systemic treatment for non-squamous NSCLC
* Negative in EGFR&ALK&ROS1
* Main organs function is normal

Exclusion Criteria:

* Have any habitus or medical history of hemorrhage, however severe it is; the patients who have non healing wounds, ulcer or fracture after any events with hemorrhage or bleeding
* Symptoms of brain metastases cannot be controlled and treated within less than 21 days
* Have participated in other clinical trials of anti-tumor medicine within 4 weeks
* Get any severe diseases or the ones that cannot be controlled

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2018-11-26 (Estimated); Primary Completion 2019-11-26 (Estimated); Study Completion 2020-11-26 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients alive and progression free at 6 months (APF6) | Estimated to be from baseline up to 2 years
  the number (%) of patients who are alive and progression free per RECIST 1.1 at 6 months after randomization per Kaplan-Meier estimate of progression free survival at 6 months.

SECONDARY OUTCOMES:
Progression Free Survival(PFS) | Estimated to be from baseline up to 2 years
  the time from randomization until the date of objective disease progression (RECIST 1.1) or death (by any cause in the absence of progression)
Overall Survival(OS) | Estimated to be from baseline up to 2 years
  the time from randomization to death from any cause
Disease Control Rate(DCR) | Estimated to be from baseline up to 2 years
  the total proportion of patients who demonstrate a response(complete responses + partial responses + stable disease ) to treatment
Objective Response Rate(ORR) | Estimated to be from baseline up to 2 years
  the total proportion of patients who demonstrate a response(complete responses + partial responses) to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chest Hospital, Beijing, Beijing Municipality, China